CLINICAL TRIAL: NCT02414659
Title: Effects of In-utero Cord Blood Collection on Post-operative Hemoglobin Levels
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Middle East Technical University (Other)
Responsible Party: Principal Investigator, Erkan Kalafat, Research Assistant, Ankara University
Other Study IDs: 003
Record Dates: First submitted 2015-04-05; First posted 2015-04-13 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Cord Blood Collection; Cesarean

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cesarean delivery, cord blood collected: Cesarean delivery patient who opted for cord blood collection during procedure. Cord blood was collected in-utero after delivery and after clamping of the umbilical cord. After cord blood collection operation was continued.
  Interventions: Procedure: Umbilical cord blood collection, in-utero
- Cesarean delivery, control: Routine cesarean delivery patients.

INTERVENTIONS:
Procedure: Umbilical cord blood collection, in-utero — Umbilical cord blood was collected during cesarean, after delivery of the baby and after clamping of the cord. Blood was collected into a standard blood donation bag with (Capacity: 450 mL) a 16 G venipuncture needle. Needle was left in place after umbilical vein is collapsed and no more blood flow happens spontaneously.
  Groups: Cesarean delivery, cord blood collected

SUMMARY:
Umbilical cord blood (UCB) collection and storage is a rapidly advancing field in hematology due to UCB's use for treatment of many hematological diseases, including but not limited to, Fanconi anemia, thalassemia, leukaemia and metabolic storage diseases. Primarily, there are two ways for UCB harvesting, first in-utero collection and second ex-utero collection. Depending on the amount of UCB collected, in-utero harvesting practice prolongs the operative time of cesarean delivery and speculatively increases intraoperative blood loss. The aim of this study is to determine UCB collection's effect on intraoperative bleeding in women undergoing elective cesarean delivery.

DETAILED DESCRIPTION:
Elective cesarean deliveries that occurred in Ankara University Department of Obstetrics and Gynecology between March 2014 and February 2015 were enrolled in the study. Deliveries were divided into two groups depending whether cord blood was collected or not. All cesarean deliveries were performed via Joel-Cohen incisions. Cord blood was harvested in-utero, i.e. while leaving the placenta inside the uterus, after delivery of the baby and clamping of the cord. After UCB collection, placenta was delivered and hysterotomy site was repaired in one layer with continuous locking. Postpartum hemorrhage prophylaxis were performed with one dose of 0.2 mg methylergonovine maleate. Postoperatively patients were hydrated with 100cc per hour infusion of isotonic liquids and bloods were drawn at eight hours postoperatively for control blood counts. Amount of blood loss was estimated by subtracting preoperative hemoglobin and hematocrit levels from postoperative hemoglobin and hematocrit. Delta hemoglobin and hematocrit levels were compared between two groups. Correlation between amount of UCB collected and blood loss was also analysed.

Patients without a preoperative blood count within 30 days prior to delivery were excluded from the study, along with patients with history of bleeding 30 days prior to delivery. Emergent cesarean deliveries, postpartum bleeding due to uterine atony, retained placenta, cesarean deliveries performed due to placental adhesion abnormalities (placenta previa, placenta accreta), patients on anticoagulation regimens (aspirin, low molecular weight heparin, heparin), patients with a post-operative haemoglobin level higher than pre-operative levels were all excluded from the study. Patients were selected at random from birth register by two people who are blind to pre and post-operative blood count results.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean deliveries
* Women with a blood count results maximum 30 days prior to delivery

Exclusion Criteria:

* Emergent cesarean deliveries
* Cesarean deliveries due to placental adhesion abnormalities or placenta previa
* Patients on anticoagulation regimens
* Postpartum bleeding due to uterine atony, retained placenta
* Patients with a history of bleeding 30 days prior to delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Elective cesarean deliveries
Sampling Method: Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Postoperative hemoglobin levels | 8 hours
  Bloods were drawn from patients during their 8th postoperative hour for control blood counts.
Postoperative hematocrit levels | 8 hours
  Bloods were drawn from patients during their 8th postoperative hour for control blood counts.

CONTACTS AND LOCATIONS:
Overall Officials: Erkan Kalafat, Principal Investigator — Department of Obstetrics and Gynecology, Ankara University Faculty of Medicine
Locations (1):
- Ankara University Faculty of Medicine, Department of Obstetrics and Gynecology, Ankara, Turkey (Türkiye)